CLINICAL TRIAL: NCT04657991
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND STUDY OF ENCORAFENIB AND BINIMETINIB PLUS PEMBROLIZUMAB VERSUS PLACEBO PLUS PEMBROLIZUMAB IN PARTICIPANTS WITH BRAF V600E/K MUTATION-POSITIVE METASTATIC OR UNRESECTABLE LOCALLY ADVANCED MELANOMA
Brief Title: A Clinical Trial of Three Study Medicines (Encorafenib, Binimetinib, and Pembrolizumab) in Patients With Advanced or Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4221016; KEYNOTE-B80 (Other: Alias Study Number); 2024-512038-13-00 (Registry Identifier: CTIS (EU)); STARBOARD (Other: Alias Study Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
Keywords: BRAF V600E/K Melanoma; BRAF; Melanoma; Advanced Melanoma; Metastatic Melanoma; Skin Cancer; Advanced Skin Cancer; Starboard; Stage 3 Melanoma; Stage 4 Melanoma; BRAF Melanoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — encorafenib; binimetinib; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Triplet Arm (Experimental): Encorafenib and Binimetinib in combination with Pembrolizumab
  Interventions: Drug: Encorafenib; Drug: Binimetinib; Drug: Pembrolizumab
- Control Arm (Active Comparator): Pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Encorafenib — Encorafenib
  Other Names: BRAFTOVI
  Arms: Triplet Arm
Drug: Binimetinib — Binimetinib
  Other Names: MEKTOVI
  Arms: Triplet Arm
Drug: Pembrolizumab — Pembrolizumab
  Other Names: KEYTRUDA

SUMMARY:
The purpose of this study is to learn about the effects of three study medicines (encorafenib, binimetinib, and pembrolizumab) given together for the treatment of melanoma that:

* is advanced or metastatic (spread to other parts of the body);
* has a certain type of abnormal gene called "BRAF"; and
* has not received prior treatment.

All participants in this study will receive pembrolizumab at the study clinic once every 3 weeks as an intravenous (IV) infusion (given directly into a vein). In addition, half of the participants will take encorafenib and binimetinib orally (by mouth) at home every day.

Participants may receive pembrolizumab for up to two years. Those participants taking encorafenib and binimetinib can continue until their melanoma is no longer responding. The study team will monitor how each participant is doing with the study treatment during regular visits at the study clinic.

DETAILED DESCRIPTION:
This study will compare the efficacy, safety, and tolerability of encorafenib and binimetinib plus pembrolizumab (Triplet Arm) versus placebo plus pembrolizumab (Control Arm) in participants with metastatic or unresectable locally advanced BRAF V600E/K mutation-positive melanoma. The study will have an open-label safety lead-in (SLI) phase to determine the safety recommend Phase 3 dose (RP3D) and pharmacokinetics (PK) of encorafenib and binimetinib plus pembrolizumab combination therapy prior to initiation of the randomized Phase 3 part of the study. Two dose levels of encorafenib in combination with binimetinib plus pembrolizumab will be explored in parallel. A minimum of 12 evaluable participants will be enrolled per dose level. During the double-blind randomized Phase 3 part of the study, approximately 216 eligible participants will be randomized in a 1:1 ratio to the Triplet Arm (at RP3D determined in the SLI) or Control Arm (approximately 108 participants per arm). Randomization will be stratified by prior systemic adjuvant therapy and stage of disease by AJCC (ED8).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥ 18 years at the time of informed consent.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Histologically confirmed unresectable (Stage IIIB, IIIC, or IIID) or metastatic (Stage IV) cutaneous melanoma, according to the AJCC 8th edition.
* Presence of at least 1 measurable lesion as detected by radiological and/or photographic methods according to RECIST v1.1.
* ECOG performance status 0 or 1.
* Documented evidence of a BRAF V600E or V600K mutation in melanoma tumor tissue as previously determined by either PCR or NGS-based local laboratory assay (eg, US FDA-approved test, CE-marked [European conformity] in vitro diagnostic in EU countries, or equivalent), obtained during the course of normal clinical care, in a CLIA- or similarly certified laboratory.
* Submission of adequate tumor tissue (archival or newly obtained; block or slides to the sponsor central laboratory(ies) during the screening period and prior to enrollment (SLI)/randomization (Phase 3).
* Have not received prior first-line systemic therapy for metastatic or unresectable locally advanced melanoma.
* Adequate bone marrow function, hepatic and renal function.
* Capable of giving signed informed consent.

Exclusion Criteria

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study (including, but not limited to, a participant who is rapidly progressing or has clinically significant tumor related symptoms, in the judgment of the investigator).
* Mucosal or ocular melanoma.
* Diagnosis of immunodeficiency or an active autoimmune disease that required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear IgA dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Unable to swallow, retain, and absorb oral medications.
* Impairment of GI function or disease which may significantly alter the absorption of oral study intervention (eg, uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, including malabsorption syndrome secondary to prior GI surgery).
* Clinically significant cardiovascular diseases,
* History of thromboembolic or cerebrovascular events ≤ 12 weeks prior to enrollment (SLI)/randomization (Phase 3). Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (ie, massive or sub-massive) deep vein thrombosis or pulmonary emboli.
* History or current evidence of RVO or current risk factors for RVO (eg, uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* Concurrent neuromuscular disorder that is associated with the potential of elevated CK (eg, inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Current noninfectious pneumonitis or history of noninfectious pneumonitis requiring steroids, or history of radiation pnuemonitis
* Evidence of HBV or HCV infection.
* Known history of a positive test for HIV or known AIDS.
* Any active infection requiring systemic therapeutic treatment within 2 weeks prior to enrollment (SLI)/ randomization (Phase 3).
* Participants with prior or current symptomatic brain metastasis, leptomeningeal disease or other active CNS metastases.
* Concurrent or previous other malignancy within 2 years of study entry, except curatively treated basal or squamous cell skin cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, Bowen's disease and Gleason ≤ 6 prostate cancer. Participants with a history of other curatively treated cancers must be reviewed with the sponsor or designee prior to entering the study.
* Participants who previously received and subsequently discontinued encorafenib and/or binimetinib and/or anti-PD-1/-L1 due to severe toxicity.
* For participants in the SLI only: Current use or anticipated need for food or drugs that are known moderate or strong CYP3A4 inhibitors during screening and through the DLT-evaluation period
* Participant has not recovered to Grade ≤ 1 from toxic effects of prior therapy and/or complications from prior surgical intervention before enrollment (SLI)/ randomization (Phase 3).
* Receipt of protocol defined medications or treatments outside of required intervals before enrollment (SLI)/randomization (Phase 3):
* Previous administration with an investigational drug ≤ 6 months prior to enrollment (SLI)/randomization (Phase 3).
* Known sensitivity or contraindication to any component of study intervention (encorafenib, binimetinib and pembrolizumab), or their excipients.
* Pregnant, confirmed by a positive β-hCG laboratory test result, or is breastfeeding (lactating).
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Safety Lead In (SLI): Incidence of Dose Limiting Toxicities (DLTs) | First 2 Cycles of Treatment (cycles are 21 days)
  A DLT is defined as any adverse event or laboratory value that is assessed as unrelated to disease, disease progression, intercurrent illness or concomitant medications/therapies occurring within the first 2 cycles of treatment.
Phase 3: Objective Response (OR) by Blinded Independent Central Review (BICR) | Time from the date of randomization until documented PD, start of subsequent anticancer therapy, or death due to any cause (approximately every 9 weeks).
  OR is defined as confirmed Best Overall response (BOR) of either CR or PR as determined by BICR assessment per RECIST 1.1

SECONDARY OUTCOMES:
Safety Lead in (SLI) and Phase 3: Incidence and severity of Adverse Events (AEs) and changes in clinical laboratory parameters, vital signs, and cardiac assessments. | Time from first dose of study intervention through 28 days after the last dose of study intervention.
  AEs, laboratory parameters, vital signs and cardiac abnormalities will be graded according to the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 4.03).
Safety Lead in (SLI) and Phase 3: Objective Response (OR) | Time from the date after the first dose of first dose (SLI) or the date of randomization (Phase 3) until documented PD, or start of subsequent anticancer therapy (approximately every 9 weeks).
  OR is defined as confirmed Best Overall Response (BOR) of either CR or PR as determined by investigator assessment per RECIST v1.1
Safety Lead in (SLI) and Phase 3: Disease Control (DC) | Time from the date after the first dose of first dose (SLI) or the date of randomization (Phase 3) until documented PD, or start of subsequent anticancer therapy (approximately every 9 weeks)
  DC is defined as confirmed BOR of CR, PR or SD, as determined by BICR and investigator assessment per RECIST v1.1.
Safety Lead in (SLI) and Phase 3: Time to Response (TTR) | Time from the date of randomization to the date of first documented response (CR or PR), as determined by investigator assessment per RECIST v1 (approximately every 9 weeks)
  TTR is defined as the time from the date of randomization to the date of first documented response (CR or PR), as determined by BICR and investigator or assessment per RECIST v1.1.
Phase 3: Overall Survival (OS) | Time from the date of randomization to the date of death due to any cause.
  OS is defined as the time from the date of randomization to the date of death due to any cause
Safety Lead In (SLI) and Phase 3: Progression Free Survival (PFS) by Investigator and BICR assessment | The time from the date of randomization to the date of first documented disease progression, as determined by investigator and BICR assessment per RECIST v1.1, or death due to any cause, whichever occurs first (approximately every 9 weeks)
  PFS by investigator is defined as the time from the date of randomization to the first date of documented disease progression as determined by investigator and BICR assessment per RECIST 1.1 or death due to any cause, whichever occurs first.
Phase 3: Duration of Response (DOR) | Time from date of first documented response (CR or PR) to the date of first documented disease progression, as determined by BICR and investigator assessment per RECIST v1.1, or death due to any cause, whichever occurs first (approximately every 9 weeks)
  DOR is defined as the time from the date of first documented response to the date of first documented disease progression, as determined by BICR and investigator assessment or death due to any cause, whichever occurs first.
Safety Lead in (SLI): Plasma concentration-time profiles and Pharmacokinetic (PK) parameter estimates for encorafenib and binimetinib. | Cycle 2, Day 1
  To measure plasma concentrations of encorafenib and its metabolite (LHY746), and binimetinib and its metabolite (AR00426032)
Phase 3: Plasma concentrations of encorafenib and binimetinib. | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1 (Each Cycle is 21 days)
  To measure the plasma concentrations of encorafenib and its metabolite (LHY746), and binimetinib and its metabolite (AR00426032)
Phase 3: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30): change from baseline in the global health status/QoL score. | Day 1 of every 3 cycles: C4D1, C7D1, C10D1, etc. for the first 24 months and then Day 1 of every 4 cycles after 24 months
  EORTC QLQ-30 includes 5 functional scales (physical, role, emotional, cognitive and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/Quality of Life scale
Phase 3: Change from baseline in Functional Assessment of Cancer Therapy-Melanoma (FACT-M) subscale score. | Day 1 of every 3 cycles: C4D1, C7D1, C10D1, etc. for the first 24 months and then Day 1 of every 4 cycles after 24 months
  The FACT-M is a melanoma-specific quality of life questionnaire that is composed of items from the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire, melanoma-specific items, and items related to melanoma surgery
Phase 3: Change from baseline in 5-level EuroQol-5D (EQ-5D-5L) index score and visual analog scale (VAS) | Day 1 of every 3 cycles: C4D1, C7D1, C10D1, etc. for the first 24 months and then Day 1 of every 4 cycles after 24 months
  The EQ-5D-5L is a standardized measure of health utility that provides a single index value of health status and contains 1 item for each of 5 dimensions of HRQoL (ie, mobility, self-care, usual activities, pain or discomfort, and anxiety or depression).
Phase 3: Change from baseline in Patient Global Impression of Severity (PGIS) score | Day 1 of every 3 cycles: C4D1, C7D1, C10D1, etc. for the first 24 months and then Day 1 of every 4 cycles after 24 months
  The PGIS is a single 1-item questionnaire designed to assess participant's overall impression of disease severity at a given point in time by using a 4-point Likert scale that ranges from (1) = "none (no symptoms)" to (4) = "severe".
Phase 3: Patient Global Impression of Change (PGIC) score | Day 1 of every 3 cycles: C4D1, C7D1, C10D1, etc. for the first 24 months and then Day 1 of every 4 cycles after 24 months
  The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change since starting treatment as rated on a 5-point Likert scale anchored by (1) "much better" to (5) "much worse", with (4) = "no change"

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (132):
- United States (14):
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - AdventHealth Orlando, Investigational Drug Services, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - The University of Kansas Cancer Center, Investigational Drug Services, Westwood, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc (OCB), Boston, Massachusetts
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Cincinnati Medical Center, West Chester, Ohio
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
- Argentina (2):
  - Instituto Alexander Fleming, CABA, Buenos Aires
  - Clinica Viedma S. A, Viedma, Río Negro Province
- Medizinische Universität Graz, Graz, Austria
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- Brazil (7):
  - Instituto de Oncologia do Paraná - IOP Matriz Mateus Leme, Curitiba, Paraná
  - Instituto de Oncologia do Paraná - IOP Oncoville, Curitiba, Paraná
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clínicas de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital Sírio-Libanês - Unidade Bela Vista, São Paulo
- Bulgaria (4):
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Medical Center Nadezhda Clinical EOOD, Sofia
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - Umhato Ead, Sofia
- CIUSSS du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec, Canada
- Czechia (3):
  - Olomouc University Hospital, Olomouc, Olomoucký kraj
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Fakultni nemocnice Bulovka, Praha 8-Liben
- Finland (2):
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki
- France (4):
  - CHU d'Amiens - Hôpital Nord, Amiens
  - CHU Grenoble Alpes, La Tronche
  - Hôpital Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
- Germany (21):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Klinik und Poliklinik für Dermatologie und Allergologie, München, Bavaria
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - SRH Wald-Klinikum Gera, Gera, Thuringia
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitätsklinikum Essen (AöR), Essen
  - Universitaetsklinikum Halle - Universitaetsklinik und Poliklinik fuer Dermatologie und Venerologie, Halle
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - University Hospital Muenster, Münster
  - Fachklinik Hornheide, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Universitätsklinikum Regensburg, Regensburg
- Greece (2):
  - General Hospital of Athens "Laiko", Athens, Attikí
  - Laiko Hospital, Athens, Attikí
- Hungary (6):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház, Szolnok, Jász-Nagykun-Szolnok
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Israel (2):
  - Soroka University Medical Center, Beersheba
  - Hadassah Medical Organization, Hadassah Medical Center, Ein-Karem, Jerusalem
- Italy (12):
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, Friuli Venezia Giulia
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Dermopatico dell'Immacolata (IDI-IRCCS), Roma, RM
  - A.O.U.S. Policlinico "Le Scotte", Siena, SI
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Istituto Tumori Giovanni Paolo II, Bari
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Istituto Oncologico Veneto IOV - IRCCS, Padua
  - AO di Perugia - Ospedale S. Maria della Misericordia, S.C Oncologia Medica, Perugia
  - Istituto Nazionale Tumori Regina Elena, Roma
- Mexico (5):
  - Preparaciones Oncológicas S.C., León, Guanajuato
  - ONCARE Viaducto Nápoles, Benito Juárez, Mexico City
  - I Can Oncology Center S.A. de C.V., Monterrey, Nuevo León
  - BRCR Global Mexico - CDMX, Mexico City
  - El Cielo Medical Center RSB, S.C, Puebla City
- Palmerston North Hospital, Palmerston North, Manawatu, New Zealand
- Oslo universitetssykehus, Radiumhospitalet, Oslo, Norway
- Poland (3):
  - Jagiellońskie Centrum Innowacji Sp. z o .o., Krakow
  - Szpital Kliniczny im. Heliodora Święcickiego UM w Poznaniu, Poznan
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
- Russia (4):
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - Ars Medika Center, LLC, Kaliningrad
  - BIH of Omsk Region "Clinical Oncological Dispensary", Omsk
  - Eurocityclinic LLC, Saint Petersburg
- Slovakia (5):
  - Onkologicky ustav sv. Alzbety, s.r.o., Bratislava
  - Narodny onkologicky ustav, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
  - Nemocnica na okraji mesta, n.o., Partizánske
  - POKO Poprad, s.r.o., Poprad
- South Africa (4):
  - WCR Office, Johannesburg, Gauteng
  - Wits Clinical Research, Johannesburg, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd, Johannesburg, Gauteng
  - Drs Alberts, Bouwer and Jordaan Inc., Pretoria, Gauteng
- Spain (17):
  - ICO-Badalona Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - CHUAC-Hospital Teresa Herrera, A Coruña
  - Hospital Universitari Vall D'Hebron, Servicio de Oncología Médica, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario de Malaga - Hospital Civil, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- UniversitätsSpital Zürich, Zürich Flughafen, Switzerland
- Turkey (Türkiye) (3):
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Istanbul, İ̇stanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul, İ̇stanbul
  - Memorial Ankara Hastanesi, Ankara
- Ukraine (4):
  - CNI KRC "Regional Cardiology Centre", Kharkiv
  - National Cancer Institute, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council "Lviv Oncological Regional Therapeutical, Lviv
  - Derzhavna ustanova Instytut zahalnoi ta nevidkladnoi khirurhii im.V.T.Zaitseva Natsionalnoi akademii, M. Kharkiv
- United Kingdom (2):
  - St. Bartholomew's Hospital, Barts Health NHS Trust, London
  - The South West Wales Cancer Institute, Swansea Bay University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schadendorf D, Dummer R, Robert C, Ribas A, Sullivan RJ, Panella T, McKean M, Santos ES, Brill K, Polli A, Pietro AD, Ascierto PA. STARBOARD: encorafenib + binimetinib + pembrolizumab for first-line metastatic/unresectable BRAF V600-mutant melanoma. Future Oncol. 2022 Jun;18(17):2041-2051. doi: 10.2217/fon-2021-1486. Epub 2022 Mar 11. PMID 35272485
- [Derived] Zimmer L, Livingstone E, Krackhardt A, Schultz ES, Goppner D, Assaf C, Trebing D, Stelter K, Windemuth-Kieselbach C, Ugurel S, Schadendorf D. Encorafenib, binimetinib plus pembrolizumab triplet therapy in patients with advanced BRAFV600 mutant melanoma: safety and tolerability results from the phase I IMMU-TARGET trial. Eur J Cancer. 2021 Nov;158:72-84. doi: 10.1016/j.ejca.2021.09.011. Epub 2021 Oct 13. PMID 34655839
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4221016